CLINICAL TRIAL: NCT04841642
Title: Feasibility and Impact of a Tele-rehabilitation Program in Patients With Chronic and Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Doctor of Health Sciences, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/50
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Chronic Non-specific Neck Pain
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy and a telerehabilitation program (Experimental): In the experimental group, an intervention based on manual therapy and a telerehabilitation program based on exercises will be carried out.
  The investigators will apply manual therapy for ten minutes a week based on cervical mobilizations and suboccipital inhibitions.
  The access to telerehabilitation will be through a web page, through which patients could see explanatory videos of the exercises as many times as they need.
  Interventions: Other: MANUAL THERAPY; Other: THERAPEUTIC EXERCISE
- Manual therapy and recommendations for home exercises (Active Comparator): In the control group, the same manual therapy intervention and recommendations for home exercises will be applied.
  This exercises recommendations will be based on a simulation of the exercise in the same session of the manual therapy of each week.
  Interventions: Other: MANUAL THERAPY; Other: THERAPEUTIC EXERCISE

INTERVENTIONS:
Other: MANUAL THERAPY — The investigators will apply manual therapy for ten minutes a week, for 8 weeks, based on cervical mobilizations and suboccipital inhibitions.
Other: THERAPEUTIC EXERCISE — The exercises recommendations will be based on a simulation of the exercises in the same session of the manual therapy of each week, helped by the physiotherapist.
  The access to telerehabilitation will be through a web page, through which patients could see explanatory videos of the exercises as many times as they need.

SUMMARY:
Chronic neck pain has a high prevalence in developed countries, being one of the main causes of years lived with disability and deterioration of the quality of life. Telerehabilitation is presented as a resource capable of favoring, with its development and implementation, the transition to a universal and quality health service. The main objective of the study is to assess the change in disability produced by a telerehabilitation program (applied in the intervention group) in patients with chronic and nonspecific neck pain compared to the recommendation of home exercises (control group).

The study that will be carried out will be a controlled and randomized clinical trial (ECCA), single-blind, longitudinal and prospective with two groups (intervention group and control group). The main study variables that are intended to be analyzed pre and post intervention are disability, quality of life, pain, adherence, and depression and anxiety.

The study will take place between June 2020 and May 2021 in specialized physiotherapy clinics.

ELIGIBILITY:
Inclusion Criteria:

* People between 18 and 65 years of age
* Neck pain of more than 3 months of evolution
* Access and knowledge in the use of the internet
* Complete the informed consent

Exclusion Criteria:

* Previous trauma to the cervical region (such as whiplash)
* Neck surgery
* Osteoporosis
* Arthritis
* Cervical radiculopathy associated with externalized cervical hernia
* Vertigo or vertebrobasilar insufficiency
* Cancer
* Vertebral fracture
* Fibromyalgia
* Cognitive impairment
* Psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in disability | Baseline, 8 weeks and 2 month after intervention.
  Using the Neck Disability Index (NDI). It is made up of 10 items and each item is scored on a 6-point Likert scale (0 to 5), leading to a total score ranging from 0 to 50 (0 to 4 = no disability; 5 to 14 = mild disability; 15 to 24 = moderate disability; 25 to 34 = severe disability; and 35 to 50 = complete disability).

SECONDARY OUTCOMES:
Changes in the health-related quality of life | Baseline, 8 weeks and 2 month after intervention.
  Using the Short Form 12 Health Survey (SF-12). It is made up of a subset of 12 items from the SF-36 (physical function, social function, physical role, emotional role, mental health, vitality, bodily pain and general health), including 1-2 items from each of the 8 scales of the SF-36.
Changes in depression and anxiety | Baseline, 8 weeks and 2 month after intervention.
  Using the Hospital Anxiety and Depression Scale (HADS). It consists of two series of seven questions (a total of 14 items), one represents the anxiety subscale and the other the depression. Each item is valued according to a four-point frequency scale that ranges from 0 to 3 (0 = I always do it; 1 = not so much; 2 = definitely not that much; 3 = not at all).
Changes in Kinesiophobia | Baseline, 8 weeks and 2 month after intervention.
  Using the Tampa Scale for Kinesiophobia-11 (TSK-11), self-report of 17 items that address fear of movement and injury relapse. Four of the items are negatively written and scored inverse (4, 8, 12 and 16). The scores are added together to obtain a total score, with higher values reflecting greater kinesiophobia.
Changes in the pain: Visual Analog Scale (VAS) | Baseline, 8 weeks and 2 month after intervention.
  Using the Visual Analog Scale (VAS). Each item is scored 0-10 (0= no pain; 10= the major pain that the patient can imagine) yielding a total between 0 and 10.
Adherence to treatment | At 4 and 8 weeks of treatment
  Using a record book of the completion of the treatment program, where the activity carried out will be reflected.
Pressure pain threshold | Baseline, 8 weeks and 2 month after intervention.
  Using a digital pressure algometer at a speed of 1 kg / cm2 / s perpendicular to the skin surface.
  The patient will be required to immediately indicate when the sensation of pressure (kg / cm2) becomes a sensation of pain, and thus terminate the compression.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, PhD, Study Director — University of Jaen
Locations (1):
- Cristina, Santa Brígida, Las Palmas, Spain